CLINICAL TRIAL: NCT03324178
Title: The Effect of Neurofeedback Training on Sustained Attention and Mind Wandering Events in Patients With Brain Injury: A Pilot Randomised Controlled Trial
Brief Title: Use of Neurofeedback to Enhance Attention After Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: Brain Injury Rehabilitation Trust (Other)
Responsible Party: Principal Investigator, Professor Jon Evans, Professor of Applied Neuropsychology, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-WS-0211
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Brain Injuries
Keywords: Neurofeedback; Attention
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: A pilot two-armed, parallel-design, individually randomised controlled trial, using stratified randomization with blocking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurofeedback training (Experimental): Sixteen 30-minute sessions of neurofeedback training performed once a day over the course of four weeks (four sessions each week)
  Interventions: Behavioral: Neurofeedback training
- Video game control group (Active Comparator): Sixteen 30-minute sessions of playing video games once a day over the course of four weeks (four sessions each week)
  Interventions: Behavioral: Video game

INTERVENTIONS:
Behavioral: Neurofeedback training — Sixteen 30-minute sessions of neurofeedback training over four weeks: 7 x 3-minute blocks of training flanked by a 3-minute resting state block with eyes-open.
  Arms: Neurofeedback training
Behavioral: Video game — Sixteen 30-minute sessions of video game playing over four weeks: 7 x 3-minute blocks flanked by a 3-minute seated relaxation.
  Arms: Video game control group

SUMMARY:
Difficulty to sustain attention over a prolonged period of time is one of the core difficulties experienced by people who have undergone traumatic brain injury. Rehabilitation of attention is often based on compensatory strategies, because of the limited impact of cognitive training on improving attentional capacity after brain injury. New therapeutic approaches to explore the plastic recovery of the brain after injury, and consequent performance improvement, are warranted.

Neurofeedback (NFB) allows the self-regulation of brain activity using visual feedback. Very recently, it has been demonstrated that NFB training targeted at reducing alpha power (alpha desynchronization NFB), can induce initial plastic changes in brain networks associated with attention. It has been proposed that NFB can improve cognitive performance by tuning oscillatory activity of the brain towards a more healthy balance between neural network flexibility and stability. It is speculated that the use of alpha desynchronization NFB training, with people who present with brain injury, can enhance sustained attention in as much as the training promotes neural variability during resting state (i.e. more flexible network configuration) and neural stability during a sustained attention task (i.e. more stable network configuration).

However, before assessing the effectiveness of the intervention, it is necessary to evaluate the feasibility and acceptability thereof. This study will recruit 14 participants and randomly assign them to two groups: a NFB group and a video games control group. Long-term changes will be evaluated at two time points for both groups: baseline and post-intervention. The NFB group will have a follow-up session one week after the intervention, to evaluate whether there are long lasting changes after NFB training. In addition, short-term changes of NFB will be evaluated for the experimental group, contrasting EEG activity immediately before and after the last NFB session.

DETAILED DESCRIPTION:
Participants taking part in the neurofeedback group will undertake sixteen 30-minute sessions of neurofeedback training, from Tuesday to Friday, distributed over the course of four weeks. Sessions will be performed at the same time each day. Each 30-min NFB session will consist of 7 x 3-minute blocks of training flanked by a 3-minute resting state block with eyes-open. During the training blocks participants will seat in front of a laptop screen displaying an image that will change according the brain activity produced by the participant. One electrode will be located at the centro parietal region of the scalp (Pz) and another one in the earlobe as a reference. Participants taking part in the control group will play video games for 30 minutes during the same number of sessions, also distributed across four weeks. The same experimental set-up will be used, but EEG activity will not be recorded. Participants will follow the same structure as the NFB group, playing video games during 7 x 3-minute blocks flanked by a 3-minute seated relaxation.

Each participant will be involved in the study for a maximum of 5 weeks. The NFB training and control sessions for all participants are expected to be completed over the course of five months.

ELIGIBILITY:
Inclusion Criteria:

* normal or corrected to normal vision
* able to provide consent
* non-progressive brain injury
* impairment of sustained attention
* stable medication regime (expected not to change during the period of the study)
* minimum computer literacy (owning a computer, laptop, tablet, ipad etc)
* native English-speakers

Exclusion Criteria:

* epilepsy
* co-morbid progressive neurological or neurodegenerative condition
* aggressive behaviour
* unhealed scalp wounds
* unable to give informed consent
* unable to cooperate with the study protocol (e.g. severe aphasia, uncorrected impairment of hearing or vision, illiteracy or unable to understand English)
* clinically unstable (e.g. due to major intercurrent illness)
* undertaking changes in the existing treatment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
Attentional performance - MAAS | Baseline and week 4
  Change in score on Mindful Attention Awareness Scale (MAAS)
  1. Mindful Attention Awareness Scale (MAAS), (Brown et al. 2003). It is a 15-item questionnaire that assesses day-to-day experiences of mind wandering.
  2. Each of the 15 questions is rated with a number between 1 to 6, with 1 being "almost always" and 6 being "almost never". The total score is calculated by averaging the answers across the 15 items. The minimum score is 1 and the maximum score is 6. The questionnaire does not have subscales.
  3. Higher scores reflect higher levels of mindfulness, this is considered to be a better outcome. Instead, lower scores reflect higher levels of mind wandering, this is considered to be a worst outcome.
  4. No subscales are combined.

SECONDARY OUTCOMES:
Attentional performance - CTET | Baseline, week 4 and week 5
  Change in score on Continuous Temporal Expectancy Task (CTET)
  1. Continuous Temporal Expectancy Task (CTET), (O'Connell 2009). It is a computerized task to evaluate sustained attention.
  2. Participants monitor a stream of stimuli to detect a low frequent target. They will be presented with 200 target trials in average, which corresponds approximately to the 10% of the total stimuli presented. 100% of target detection is the highest possible score.
  3. Higher percentage of target detection reflects better sustained attention capacity and it is considered to be a better outcome.
  4. No subscales are combined.
Attentional performance - TEA | Baseline and week 4
  Change in score on Test of Everyday Attention (TEA)
  1. Test of Every Day Attention (TEA), (Robertson et al. 1996). It is a clinical assessment of attention. In this study, only three subtests will be used that evaluate sustained attention: (1) elevator counting, (2) telephone search while counting and (3) lottery 2a. Scale range for the subtest Elevator Counting: 0 - 7. 2b. Scale Range for the subtest Telephone Search while counting: -1.0 - 17.0 (raw score).
  2c. Scale Range for the subtest Lottery: 0 - 10 (raw score) 3a. Elevator Counting: A score of 7 (maximum) is considered normal. 5 or less is considered definitely abnormal.
  3b. Telephone Search while counting: lower raw scores are considered better output 3c. Lottery: higher raw scores are considered better output. 4. The subscales will not be combined

CONTACTS AND LOCATIONS:
Overall Officials: Jon Evans, PhD, Study Director — Professor of Applied Neuropsychology
Locations (1):
- Brain Injury Rehabilitation Trust, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided